CLINICAL TRIAL: NCT00393471
Title: A Double-blind Study Evaluating the Efficacy and Safety of the Combination of Etanercept and Methotrexate in Comparison to Etanercept Alone or Methotrexate Alone in Rheumatoid Arthritis Patients.
Brief Title: Study Comparing Etanercept Plus Methotrexate to Either Etanercept or Methotrexate Alone in Rheumatoid Arthritis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0881A1-308
Record Dates: First submitted 2006-10-26; First posted 2006-10-27 (Estimated); Last update posted 2023-12-13 (Actual); Status verified 2006-10

CONDITIONS: Active Rheumatoid Arthritis
Keywords: Arthritis; Rheumatoid; Safety
MeSH Terms: conditions — Arthritis | interventions — Etanercept

INTERVENTIONS:
Drug: Etanercept

SUMMARY:
To compare the therapeutic and radiographic effects and safety between etanercept, methotrexate, and the etanercept/methotrexate combination in patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
Etanercept is an injection administered under the skin twice weekly. Methotrexate is a tablet to be taken once weekly. Patients will not know which treatment they are on. Patients will need to meet the study criteria to be enrolled in the study and sign an informed consent.

ELIGIBILITY:
Inclusion:

- Generally healthy of at least 18 years of age with active rheumatoid arthritis.

Exclusion:

- A history or presence of clinically important medical disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 615
Dates: Start 2000-10; Study Completion 2001-10

PRIMARY OUTCOMES:
The objective of this study is to evaluate the therapeutic response including radiographic changes and safety of etanercept alone, methotrexate (MTX) alone, and the combination of etanercept and MTX in patients with rheumatoid arthritis (RA)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Australia, medinfo@wyeth.com; Trial Manager, Principal Investigator — For Austria, WPVIMED@wyeth.com; Trial Manager, Principal Investigator — For Belgium, trials-BEL@wyeth.com; Trial Manager, Principal Investigator — For Czech Republic, WPPGCLI@wyeth.com; Trial Manager, Principal Investigator — For Denmark, Finland, Norway, and Sweden, medinfonord@wyeth.com; Trial Manager, Principal Investigator — For France, infomedfrance@wyeth.com; Trial Manager, Principal Investigator — For Germany, medinfoDEU@wyeth.com; Trial Manager, Principal Investigator — For Greece, decresg@wyeth.com; Trial Manager, Principal Investigator — For Italy, descresg@wyeth.com; Trial Manager, Principal Investigator — For Netherlands, trials-NL@wyeth.com; Trial Manager, Principal Investigator — For Poland, WPWZMED@wyeth.com; Trial Manager, Principal Investigator — For Romania, WVPIMED@wyeth.com; Trial Manager, Principal Investigator — For Spain, infomed@wyeth.com; Trial Manager, Principal Investigator — For UK/Great Britian, ukmedinfo@wyeth.com
Locations (82):
- Australia (3):
  - St Leonards, New South Wales
  - Adelaide
  - Southport
- Vienna, Austria
- Belgium (5):
  - Brussels
  - Diepenbeek
  - Ghent
  - Leuven
  - Liège
- Czechia (4):
  - Česká Lípa
  - Prague
  - Terezín
  - Zlín
- Denmark (2):
  - Copenhagen
  - Herlev
- Finland (4):
  - Kuopio
  - Rauma
  - Tampere
  - Vantaa
- France (11):
  - Bordeaux
  - Brest
  - Créteil
  - Grenoble
  - Le Kremlin-Bicêtre
  - Montpellier
  - Nice
  - Paris
  - Rouen
  - Strasbourg
  - Toulouse
- Germany (9):
  - Berlin
  - Cologne
  - Erlangen
  - Herne
  - Leipzig
  - München
  - Plauen
  - Vogelsang
  - Würzburg
- Greece (2):
  - Athens
  - Thessaloniki
- Israel (2):
  - Jerusalem
  - Petah Tikva
- Italy (7):
  - Ferrara
  - Florence
  - Genova
  - Milan
  - Napoli
  - Pavia
  - Udine
- Netherlands (9):
  - Alkmaar
  - Arnhem
  - Doetinchem
  - Enschede
  - Leeuwarden
  - Maastricht
  - Nijmegen
  - Tilburg
  - Venlo
- Norway (2):
  - Drammen
  - Oslo
- Poland (5):
  - Elblag
  - Kalisz
  - Krakow
  - Warsaw
  - Wroclaw
- Lisbon, Portugal
- Romania (2):
  - Bucharest
  - Cluj-Japoca
- Spain (5):
  - Barcelona
  - Guadalajara
  - Madrid
  - Santander
  - Santiago de Compostela
- Sweden (5):
  - Jönköping
  - Kalmar
  - Linköping
  - Stockholm
  - Uppsala
- United Kingdom (3):
  - London
  - North Yorks
  - Trent

REFERENCES:
- [Derived] Gallo G, Brock F, Kerkmann U, Kola B, Huizinga TW. Efficacy of etanercept in combination with methotrexate in moderate-to-severe rheumatoid arthritis is not dependent on methotrexate dosage. RMD Open. 2016 Apr 21;2(1):e000186. doi: 10.1136/rmdopen-2015-000186. eCollection 2016. PMID 27175292
- [Derived] van der Heijde D, Klareskog L, Landewe R, Bruyn GA, Cantagrel A, Durez P, Herrero-Beaumont G, Molad Y, Codreanu C, Valentini G, Zahora R, Pedersen R, MacPeek D, Wajdula J, Fatenejad S. Disease remission and sustained halting of radiographic progression with combination etanercept and methotrexate in patients with rheumatoid arthritis. Arthritis Rheum. 2007 Dec;56(12):3928-39. doi: 10.1002/art.23141. PMID 18050208